CLINICAL TRIAL: NCT06593912
Title: Comprehensive Assessment of Peroneal Tendon Injuries - Evaluation and Treatment
Brief Title: Functional and Patient-reported Outcome After Peroneal Tendon Surgery and Different Immobilization Protocols
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Capio Group (Other); ATLEVA Fotcenter (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAPTI
Record Dates: First submitted 2024-09-03; First posted 2024-09-19 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Tendon Tear; Tendon Rupture; Tendon Injuries; Surgery
MeSH Terms: conditions — Tendon Injuries | interventions — AIEOP acute lymphoblastic leukemia protocol

STUDY DESIGN:
Intervention Model Description: Randomized controlled study comparing two different immobilization protocols.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cast (Active Comparator): Postoperative immobilization with cast in 6 weeks.
  Interventions: Procedure: Standard protocol
- Cast + Air Stirrup (Active Comparator): Postoperative immobilization with cast in 3 weeks followed by Air Stirrup in 3 weeks. Early range of motion after 3 weeks postoperative.
  Interventions: Procedure: Early Functional Training

INTERVENTIONS:
Procedure: Early Functional Training — Early functional training after 3 weeks using Air Stirrup compared to cast (standard protocol) after peroneal tendon surgery.
  Arms: Cast + Air Stirrup
Procedure: Standard protocol — Cast 6 weeks after peroneal tendon surgery (standard protocol)
  Arms: Cast

SUMMARY:
Patients with surgery of a peroneal tendon injury in Gothenburg, Sweden, will be randomized to one of two different postoperative protocols. Before and after surgery the patients will perform biomechanical evaluation and also fill out questionnaires including PROMs. All evaluations will be performed on both limbs.

DETAILED DESCRIPTION:
Patients admitted for surgery because of peroneal tendon injury will be randomized to one of two postoperative immobilization protocols. In group A the patients will use a cast for 6 weeks after surgery. In group B, the patients will use a cast for 3 weeks followed by a Air Stirrup for 3 weeks. The patients in group B will start unloaded range of motion 3 weeks after surgery. Both groups are allowed to weight-bear directly after surgery. The patients will be evaluated before and several times after surgery. Patient-reported outcome measures (PROMs) will be used to evaluate changes in patient quality of life between the two interventions. A biomechanical evaluation of the ankle, knee and hip kinematics and kinetics during walking, running and walking will also be performed before and repeatedly after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Surgery of peroneal tendon rupture and/or rupture of ligament and/or rupture of retinacle

Exclusion Criteria:

* Extensive surgery needed, such as for example heel osteotomy
* Previous surgery in the affected area
* Previous injury in the healthy foot/leg that impairs function
* Neuromuscular disease
* Impaired language comprehension
* Age under 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
NRS | Preoperative and 3 weeks, 6 weeks, 3 months, 6 months, 12 months and 24 months postoperative.
  Pain will be graded using Numeric Rating Scale (NRS) ranging from 0 to 10, whereas 0 is corresponding to no pain and 10 is corresponding to the worst pain imaginable.
  Patients will be asked to select a corresponding number (0 - 10) to indicate the pain intensity they are experiencing during an average day, before taking the functional tests, during the tests and after taking the functional tests. In follow-ups that does not include any functional tests, the patients will only grade pain during an average day.

SECONDARY OUTCOMES:
Calf circumference | Preoperative and 6 months, 12 months and 24 months postoperative.
  The widest part of the calf will be measured.
Range of motion | Preoperative and postoperative at 6 weeks, 3 months, 6 months, 12 months and 24 months.
  Range of motion (ROM) will be measured with inclinometer. Patients will be barefoot. ROM will be measured preoperative and postoperative after 6 weeks, 3 months, 6 months, 12 months and 24 months.
  The first two measurements after surgery (6 weeks, 3 months) will be carried out unloaded. The subsequent measurements (6 months, 12 months, 24 months) will be carried out loaded.
Balance | Preoperative and postoperative at 6 months, 12 months and 24 months.
  The patients balance will be measured with stabilometry.
Biomechanical evaluation | Preoperative and postoperative at 6 months, 12 months and 24 months.
  A biomechanical evaluation of the ankle, knee and hip kinematics and kinetics during walking, running, and jumping will be performed before and after surgery (6 months, 12 months and 24 months). For collection of the data, 16 Qualisys 7+ cameras (Qualisys AB, Gothenburg, Sweden) and 4 force plates will be used. 55 reflectors will be attached on the patient's body to be able to detect segmental movements. Kinetic data will be evaluated in power (watt) in ankle, knee and hip. Comparison will be performed between groups and limbs in power (LSI) - injured side/healthy side *100 expressed in percent. The range in LSI is between 0-100% and the higher value, the better outcome.
Electromyography (EMG) | Preoperative and postoperative at 6 months, 12 months and 24 months.
  EMG electrodes on the medial and lateral Gastrocnemius, Soleus and Tibialis Anterior, Quadriceps and trunk muscles will be attached on the patient in order to measure how the muscles are recruited during walking, running and jumping. Both healthy and injured sides will be analyzed. The electrical activity in the muscles will be evaluated. Comparison will be performed between groups and limbs in power (LSI) - injured side/healthy side * 100 expressed in percent. The range in LSI is between 0-100% and the higher value, the better outcome.
Cutting test | Preoperative and postoperative at 6 months, 12 months and 24 months.
  Cutting test will be performed according to standard module.
Heel-rise work test | Preoperative and postoperative at 6 months, 12 months and 24 months.
  Ankle plantar flexion endurance and heel-rise height will be evaluated using MuscleLab® during a heel-rise work test.
Background questions | Preoperative and 3 weeks, 6 weeks, 3 months, 6 months, 12 months and 24 months postoperative.
  During all follow-ups (including preoperative) the patients will fill out questionnaires. The questionnaires contain questions concerning, for example, fear of physical activity, fear of re-injuring oneself, satisfaction with the treatment, whether they have experienced complications, time on sick leave, etc.
The Self-Reported Foot and Ankle Score (SEFAS) | Preoperative and postoperative at 6 months, 12 months and 24 months.
  SEFAS is a questionnaire designed to evaluate disorders of the foot and ankle.
  The score covers different constructs that are not reported separately in subscales: pain, function including limitations of function, and other symptoms. Each of the 12 multiple-choice questions is scored from 0 to 4; thus, 0 total points represents the most severe disability and 48 represents normal function.
Foot and Ankle Outcome Score (FAOS) | Preoperative and postoperative at 6 months, 12 months and 24 months.
  The FAOS is a patient-reported foot- and ankle-specific questionnaire including 42 items in 5 subscales evaluating pain, symptoms, function of daily living (ADL), function in sport and recreation, and quality of life (QOL). Standardized answer options are provided, and each question is rated on a scale from 0 to 4. A score is calculated for each subscale after which raw scores for each subscale are transformed to a scale ranging from 0 to 100 and presented graphically as the FAOS profile. The minimum possible total score for each subscale is 0 points, a condition that represents the most severe disability, whereas the maximum of 100 points represents normal ankle function.
Physical Activity Scale (PAS) | Preoperative and postoperative at 6 months, 12 months and 24 months.
  Physical activity questionnaire. A patient reported outcome used fot the purpose to evaluate the patients self estimated physical activity level. The scale is from 1 to 6 and the higher score, the better outcome.
EuroQol- 5 Dimension (EQ-5D) | Preoperative and postoperative at 6 months, 12 months and 24 months.
  Descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has three levels: no problems, some problems, and extreme problems. The EQ-5D index is a weighted total value of the score that is calculated after being adjusted for cultural differences.
  The answers given to EQ-5D permit to find 243 unique health states or can be converted into EQ- 5D index an utility scores anchored at 0 for death and 1 for perfect health.

CONTACTS AND LOCATIONS:
Overall Officials: Katarina Nilsson Helander, Ass prof, Principal Investigator — Sahlgrenska University Hospital/Gothenburg University
Locations (1):
- Department of Orthopedics, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No